CLINICAL TRIAL: NCT04055987
Title: The Use of Electropalatography to Improve Speech Sound Production in Deaf Adults With Cochlear Implants
Brief Title: Use of Electropalatography to Improve Speech Sound Production
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI retired and co investigator left institution.
Sponsor: Molloy College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04190121
Record Dates: First submitted 2019-04-22; First posted 2019-08-14 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss | interventions — Models, Biological

STUDY DESIGN:
Intervention Model Description: Two groups of hearing-impaired persons with cochlear implants.One group will have congenital hearing loss. The second group will include individuals with acquired hearing loss.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Congenitally deaf (Experimental): Prior and post speech training, participants will read aloud a standard paragraph (Rainbow passage), complete a traditional speech test (Goldman Fristoe Test of Articulation - 3) to assess the sounds of the English language in all word positions (initial, medial, final) and read a list of consonant-vowel-consonant (CVC) combinations. Individual treatment will be provided once a week for 10 consecutive weeks. Traditional speech intervention with visual biofeedback from the EPG will be used. Auditory feedback will be provided through the participants own cochlear implant.
  Interventions: Behavioral: Visual biofeedback, auditory feedback and models
- Adventitiously deaf (Experimental): Prior and post speech training, participants will read aloud a standard paragraph (Rainbow passage), complete a traditional speech test (Goldman Fristoe Test of Articulation - 3) to assess the sounds of the English language in all word positions (initial, medial, final) and read a list of CVC combinations. Individual treatment will be provided once a week for 10 consecutive weeks. Traditional speech intervention with visual biofeedback from the EPG will be used. Auditory feedback will be provided through the participants own cochlear implant.
  Interventions: Behavioral: Visual biofeedback, auditory feedback and models

INTERVENTIONS:
Behavioral: Visual biofeedback, auditory feedback and models — The EPG software program allows the speech clinician to model and comment upon the visual patterns during tongue/palate contact and to replay the participant's production for additional correction or reinforcement productions. Auditory feedback will be used to facilitate participant's perception of differences in production.

SUMMARY:
The purpose of this proposed study is to examine the benefits of using electropalatography (EPG) during speech therapy with adult individuals who are either congenitally deaf or adventitiously deaf and use a cochlear implant.

DETAILED DESCRIPTION:
It has been established in numerous research studies that there is a definitive link between speech perception and speech production, in that what one can perceive, one can produce. Hearing loss disrupts this link and while cochlear implants make a significant difference in perception of sound, adults who are deaf and receive a cochlear implant (CI) do not gain the same perceptual benefits as children who are deaf and are implanted at a young age. Thus, the speech production of the adult CI user is reported to be less intelligible. The purpose of this proposed study is to examine the benefits of using electropalatography (EPG) during speech therapy with adult individuals who are either congenitally deaf or adventitiously deaf and use a cochlear implant. The investigators have proposed to study 10 CI users (5 in each etiological group) who will undergo speech intelligibility testing, and receive speech therapy (1x/week for 10 weeks) using EPG that provides both visual (biofeedback) and auditory feedback. It is hypothesized that the biofeedback in addition to the auditory feedback from the CI will result in an increase in articulation skills and thus the speech intelligibility in these individuals will improve significantly.

ELIGIBILITY:
Inclusion Criteria:

* All participants in this study will be at least 3 years post-implant and they must use the implants consistently.
* Participants who have adventitious/acquired hearing loss must have had normal hearing through their 18th year.
* Participants with congenital hearing loss will have received oral or total communication education, worn hearing aids and consider themselves to be "oral deaf" adults.

Exclusion Criteria:

* Individuals who do not meet this criteria will be excluded from the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Improved Speech Intelligibility | 10 weeks.
  Change from baseline in speech intelligibility within a 10 week period after exposed to visual display of speech sound production.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Saulle, Ph.D, Principal Investigator — Molloy College; Nancy McGarr, Ph.D., Principal Investigator — Molloy College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernhardt, B. H., Loyst, D., Pichora-Fuller, K., & Williams, R. (2000). Speech production outcomes before and after palotometry for a child with a cochlear implant. Journal-Academy of Rehabilitative Audiology, 33, 11-38.
- [Background] Bernhardt B, Gick B, Bacsfalvi P, Ashdown J. Speech habilitation of hard of hearing adolescents using electropalatography and ultrasound as evaluated by trained listeners. Clin Linguist Phon. 2003 Apr-May;17(3):199-216. doi: 10.1080/0269920031000071451. PMID 12858839
- [Background] Byun TM, Hitchcock ER. Investigating the use of traditional and spectral biofeedback approaches to intervention for /r/ misarticulation. Am J Speech Lang Pathol. 2012 Aug;21(3):207-21. doi: 10.1044/1058-0360(2012/11-0083). Epub 2012 Mar 21. PMID 22442281
- [Background] Dagenais PA. Electropalatography in the treatment of articulation/phonological disorders. J Commun Disord. 1995 Dec;28(4):303-29. doi: 10.1016/0021-9924(95)00059-1. PMID 8576412
- [Background] Dagenais PA, Critz-Crosby P. Consonant lingual-palatal contacts produced by normal-hearing and hearing-impaired children. J Speech Hear Res. 1991 Dec;34(6):1423-35. doi: 10.1044/jshr.3406.1423. PMID 1787723
- [Background] Fabus, R., Raphael, L., Gatzonis, S., Dondorf, K., Giardina, K., Cron, S., & Badke, B. (2015). Preliminary case studies investigating the use of electropalatography (EPG) manufactured by CompleteSpeech® as a biofeedback tool in intervention. International Journal, 3(1), 11-23.
- [Background] Fletcher SG, Hasegawa A. Speech modification by a deaf child through dynamic orometric modeling and feedback. J Speech Hear Disord. 1983 May;48(2):178-85. doi: 10.1044/jshd.4802.178. PMID 6621010
- [Background] Fletcher SG, Dagenais PA, Critz-Crosby P. Teaching consonants to profoundly hearing-impaired speakers using palatometry. J Speech Hear Res. 1991 Aug;34(4):929-42. doi: 10.1044/jshr.3404.929. PMID 1956200
- [Background] Fletcher, S., Hasegawa, A., McCutcheon, M., & Gilliom, J. (1980). Use of linguapalatal contact patterns to modify articulation in a deaf adult. In D. L. McPherso (Ed.), Advances in prosthetic devices for the deaf: A technical workshop (pp.127-133). Rochester, MD: NTID Press.
- [Background] Gibbon, F., Stewart, F., Hardcastle, W. J., & Crampin, L. (1999). Widening access to electropalatography for children with persistent sound system disorders. American Journal of Speech-Language Pathology, 8(4), 319-334.
- [Background] Goldman, R., & Goldman, F. M. (2000). Fristoe Test of Articulation. American Guidance Service.
- [Background] Lane H, Perkell J, Svirsky M, Webster J. Changes in speech breathing following cochlear implant in postlingually deafened adults. J Speech Hear Res. 1991 Jun;34(3):526-33. doi: 10.1044/jshr.3403.526. PMID 2072676
- [Background] Martin, K. L., Hirson, A., Herman, R., Thomas, J., & Pring, T. (2007). The efficacy of speech intervention using electropalatography with an 18-year-old deaf client: A single case study. Advances in Speech Language Pathology, 9(1), 46- 56.
- [Background] McGarr NS. The intelligibility of deaf speech to experienced and inexperienced listeners. J Speech Hear Res. 1983 Sep;26(3):451-8. doi: 10.1044/jshr.2603.451. PMID 6645470
- [Background] McGarr, N. S., Raphael, L. J., Kolia, B., Vorperian, H. K., & Harris, K. (2004). Sibilant production in speakers who have hearing loss: Electropalatographic and perceptual evidence. The Volta Review, 104(3), 119.
- [Background] Pantelemidou V, Herman R, Thomas J. Efficacy of speech intervention using electropalatography with a cochlear implant user. Clin Linguist Phon. 2003 Jun-Aug;17(4-5):383-92. doi: 10.1080/0269920031000079958. PMID 12945614
- [Background] Parsloe R. Use of the speech pattern audiometer and the electropalatograph to explore the speech production/perception relationship in a profoundly deaf child. Int J Lang Commun Disord. 1998 Jan-Mar;33(1):109-21. doi: 10.1080/136828298247947. PMID 9673223
- [Background] Pratt, S. R. (2007). Using electropalatographic feedback to treat the speech of a child with severe-to-profound hearing loss. The Journal of Speech and Language Pathology-Applied Behavior Analysis, 2(2), 213.
- [Background] Shriberg, L. D. (1980). An intervention procedure for children with persistent /r/ errors. Language, Speech, and Hearing Services in Schools, 11(2), 102-110. SmartPalate Overview. (n.d.). Retrieved from http://completespeech.com/smartpalate/smartpalate_overview/
- [Background] Subtenly, J. D., Orlando, N. A., & Whitehead, R. L. (1981). Speech and voice characteristics of the deaf. Washington, DC: The Alexander Graham Bell Association of the Deaf.
- [Background] Waldstein RS. Effects of postlingual deafness on speech production: implications for the role of auditory feedback. J Acoust Soc Am. 1990 Nov;88(5):2099-114. doi: 10.1121/1.400107. PMID 2269726